CLINICAL TRIAL: NCT03039504
Title: Clinical Evaluation of Effectiveness and Safety of Dietary Supplement Potensa in Men With Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Center, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Potensa02-2017
Record Dates: First submitted 2017-01-23; First posted 2017-02-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Erectile Dysfunction
Keywords: Succinates; Dietary supplement
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potensa (Experimental): succinate-based dietary supplement
  Interventions: Dietary Supplement: Potensa, a succinate-based dietary supplement
- Placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Potensa, a succinate-based dietary supplement — Potensa - a dietary supplement: 4 capsules (2 white 200mg each and 2 blue 200 mg each) once a day with a meal or immediately after a meal, preferably after breakfast, for 3 months.
  Arms: Potensa
Dietary Supplement: Placebo — Placebo: 4 capsules (2 white 200mg each and 2 blue 200 mg each) once a day with a meal or immediately after a meal, preferably after breakfast, for 3 months.
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo-controlled, comparative, prospective study (clinical evaluation) of the effectiveness and safety of dietary supplement Potensa in men with mild to moderate erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Men, 18 years of age or older;
* Patients diagnosed with "erectile dysfunctions" of various pathogenesis, typical form without complications;
* Ability to read and understand informed consent in order to participate in the study;
* Ability to follow study's conditions.

Exclusion Criteria:

* Oncological illnesses, except those in complete remission for at least 5 years;
* Conditions that may require emergency or planned hospitalization in the next 6 months;
* Extragenital endocrine conditions (hormonally active) (thyroid, adrenal glands, pituitary, hypothalamus);
* Surgeries on sex organ within 1 year of the screening;
* Any surgeries within 3 months of the screening;
* Psychiatric illnesses;
* Diabetes mellitus;
* Cryptorchidism
* Taking other dietary supplements that can affect erectile dysfunction within 1 month of participating in the study;
* High risk of non-compliance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the International Index of Erectile Function (IIEF) score | Baseline - 30 days
  Self reported erectile function; higher score indicates less dysfunction
Change from baseline in the International Index of Erectile Function (IIEF) score | Baseline - 60 days
  Self reported erectile function; higher score indicates less dysfunction
Change from baseline in the International Index of Erectile Function (IIEF) score | Baseline - 90 days
  Self reported erectile function; higher score indicates less dysfunction
Change from baseline in the Aging Male Symptome Scale (AMS) score | Baseline - 30 days
  Self reported symptoms; lower score indicates fewer/lesser symptoms
Change from baseline in the Aging Male Symptome Scale (AMS) score | Baseline - 60 days
  Self reported symptoms; lower score indicates fewer/lesser symptoms
Change from baseline in the Aging Male Symptome Scale (AMS) score | Baseline - 90 days
  Self reported symptoms; lower score indicates fewer/lesser symptoms
Change from baseline in the Spielberger-Hanin anxiety test | Baseline - 30 days
  Self-administered questionnaire; higher score indicates more anxiety
Change from baseline in the Spielberger-Hanin anxiety test | Baseline - 60 days
  Self-administered questionnaire; higher score indicates more anxiety
Change from baseline in the Spielberger-Hanin anxiety test | Baseline - 90 days
  Self-administered questionnaire; higher score indicates more anxiety
Change from baseline in testosterone levels | Baseline - 30 days
  Blood testosterone levels, pg/ml
Change from baseline in testosterone levels | Baseline - 60 days
  Blood testosterone levels, pg/ml
Change from baseline in testosterone levels | Baseline - 90 days
  Blood testosterone levels, pg/ml
Change from baseline in follicle stimulating hormone (FSH) levels | Baseline - 30 days
  Blood FSH levels, mIU/ml
Change from baseline in follicle stimulating hormone (FSH) levels | Baseline - 60 days
  Blood FSH levels, mIU/ml
Change from baseline in follicle stimulating hormone (FSH) levels | Baseline - 90 days
  Blood FSH levels, mIU/ml
Change from baseline in luteinizing hormone (LH) levels | Baseline - 30 days
  Blood LH levels, mIU/ml
Change from baseline in luteinizing hormone (LH) levels | Baseline - 60 days
  Blood LH levels, mIU/ml
Change from baseline in luteinizing hormone (LH) levels | Baseline - 90 days
  Blood LH levels, mIU/ml
Change from baseline in Sex Hormone Binding Globulin (SHBG) levels | Baseline - 30 days
  Blood SHBG levels, nmol/L
Change from baseline in Sex Hormone Binding Globulin (SHBG) levels | Baseline - 60 days
  Blood SHBG levels, nmol/L
Change from baseline in Sex Hormone Binding Globulin (SHBG) levels | Baseline - 90 days
  Blood SHBG levels, nmol/L
Change from baseline in inhibin B levels | Baseline - 90 days
  Blood inhibin B levels, ng/L
Change from baseline in homocystein levels | Baseline - 90 days
  Blood homocystein levels, umol/L

SECONDARY OUTCOMES:
Quality of life | Baseline - 90 days
  Based on the results of Spielberger-Hanin anxiety test (score).
Quality of life | Baseline - 90 days
  Based on the results of International Index of Erectile Function (IIEF) test (score)
Quality of life | Baseline - 90 days
  Based on the results of Aging Male Symptoms (AMS) test (score)
Positive dynamics of the primary endpoints | 30th, 60th, 90th days
  Percent of patients corresponding to the primary endpoints with positive dynamics

CONTACTS AND LOCATIONS:
Overall Officials: Evgenii A Efremov, MD, Principal Investigator — N.A. Lopatkin Urology and Interventional Radiology Research Center
Locations (2):
- Russia (2):
  - N.A. Lopatkin Urology and Interventional Radiology Research Center, Moscow
  - Ryazan State Medical University named after academician I.P. Pavlov, Ryazan

IPD SHARING:
Plan to Share IPD: No